CLINICAL TRIAL: NCT03447964
Title: Plasma Dihydroceramides Are Associated With Hepatic Steatosis in Type 1 and Type 2 Diabetes
Acronym: CERADIAB
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Joe Elie Salem, Assistant director, clinical investigation center Paris Est, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC14-21-17-12
Record Dates: First submitted 2018-01-31; First posted 2018-02-27 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1
Keywords: sphingolipids; hepatic steatosis; non-alcoholic fatty liver disease; macrovascular complications; insulin resistance; microvasclar complications; NAFLD
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Fatty Liver; Non-alcoholic Fatty Liver Disease; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — plasma samples and dosing of Sphingolipids
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type 1 diabetes: dosing of sphingolipids
  Interventions: Other: dosing of sphingolipids
- Type 2 diabetes: Dosing of sphingolipids
  Interventions: Other: dosing of sphingolipids

INTERVENTIONS:
Other: dosing of sphingolipids — - Measuring the concentration of many species of sphingomyelins, ceramides, dihydroceramides and sphingosine

SUMMARY:
Sphingolipids are associated with metabolic diseases. Distribution of plasma sphingolipids in type 1 and type 2 diabetes has never been studied. The objective of the CERADIAB study is to compare plasma sphingoliplids concentrations in type 1 and type 2 diabetic patients.

DETAILED DESCRIPTION:
Sphingolipids represent a major class of lipids that are structural and signaling molecules. Major bioactive sphingolipids include ceramide, dihydroceramide, sphingosine, sphingosine-1-phosphate and sphingomyelin.

Sphingoliplids are involved in development of various chronic metabolic diseases. Some ceramides species are implicated in pancreatic β-cell apoptosis and in insulin resistance in muscle, fat and liver. Some studies have shown association between inhibition of ceramide synthesis, insulin sensibility and lower hepatic steatosis. The deposition of hepatic lipids, especially triacylglycerol, defines the development of hepatic steatosis. However, sphingolipids appear to play an important role in non-alcoholic fatty liver disease (NAFLD) and in its progression. Changes in plasma shingolipids concentrations may also contribute to the pathogenesis in cardiovascular disease and atherosclerosis. Distribution of plasma sphingolipids concentrations in type 1 and type 2 diabetes has poorly been studied.

The objective of the CERADIAB study is to compare plasma sphingoliplids concentrations in type 1 and type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* type 1 or 2 diabetes

Exclusion Criteria:

* atypical diabetes

  * family dyslipidemia
  * nonmetabolic hepatopathy
  * severe renal failure
  * corticosteroid or immunosuppressive therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients suffering of diabetes type 1 or type 2.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2017-09-16 (Actual); Study Completion 2017-09-16 (Actual)

PRIMARY OUTCOMES:
Comparison of plasma total ceramides concentration in type 2 diabetic patients versus type 1 diabetic patients. | Samples taken in 1 single time in the morning, patients fast for 12 hours, on 1 single day
  Three-hundred microlitres of plasma were used to quantify dihydroceramides, ceramides, sphingomyelins and sphingosine content. The lipid subspecies were extracted and analysed by Liquid Chromatography Mass Spectrometry (LC-MS/MS), at the Lipidomic Core Facility of the University of Bourgogne (Dijon, France).

SECONDARY OUTCOMES:
- Comparison of plasma total dihydroceramides concentration in type 2 diabetic patients versus type 1 diabetic patients. | Samples taken in 1 single time in the morning, patients fast for 12 hours, on 1 single day
  Three-hundred microlitres of plasma were used to quantify dihydroceramides, ceramides, sphingomyelins and sphingosine content. The lipid subspecies were extracted and analysed by Liquid Chromatography Mass Spectrometry (LC-MS/MS), at the Lipidomic Core Facility of the University of Bourgogne (Dijon, France).
- - Comparison of plasma total sphingomyelins concentration in type 2 diabetic patients versus type 1 diabetic patients. | Samples taken in 1 single time in the morning, patients fast for 12 hours, on 1 single day
  Three-hundred microlitres of plasma were used to quantify dihydroceramides, ceramides, sphingomyelins and sphingosine content. The lipid subspecies were extracted and analysed by Liquid Chromatography Mass Spectrometry (LC-MS/MS), at the Lipidomic Core Facility of the University of Bourgogne (Dijon, France).
- Comparison of plasma total sphingosine concentration in type 2 diabetic patients versus type 1 diabetic patients. | Samples taken in 1 single time in the morning, patients fast for 12 hours, on 1 single day
  Three-hundred microlitres of plasma were used to quantify dihydroceramides, ceramides, sphingomyelins and sphingosine content. The lipid subspecies were extracted and analysed by Liquid Chromatography Mass Spectrometry (LC-MS/MS), at the Lipidomic Core Facility of the University of Bourgogne (Dijon, France).
- Comparison of plasma ceramide species (C16, C18, C20, C22, C23, C24, C24:1, C26:1, C26:2 ceramides) concentration in type 2 diabetic patients versus type 1 diabetic patients. | Samples taken in 1 single time in the morning, patients fast for 12 hours, on 1 single day
  Three-hundred microlitres of plasma were used to quantify dihydroceramides, ceramides, sphingomyelins and sphingosine content. The lipid subspecies were extracted and analysed by Liquid Chromatography Mass Spectrometry (LC-MS/MS), at the Lipidomic Core Facility of the University of Bourgogne (Dijon, France).
- Comparison of plasma dihydroceramide species (C18/16, C18/18, C18/20, C18/22, C18/23, C18/24, C18/24:1, C18/26:1, C18/26:2 dihydroceramides) concentration in type 2 diabetic patients versus type 1 diabetic patients. | Samples taken in 1 single time in the morning, patients fast for 12 hours, on 1 single day
  Three-hundred microlitres of plasma were used to quantify dihydroceramides, ceramides, sphingomyelins and sphingosine content. The lipid subspecies were extracted and analysed by Liquid Chromatography Mass Spectrometry (LC-MS/MS), at the Lipidomic Core Facility of the University of Bourgogne (Dijon, France).
- Correlation between sphingolipids species concentrations and NAFLD biomarkers (steatotest, NASHtest and fibrotest) | Samples taken in 1 single time in the morning, patients fast for 12 hours, on 1 single day
  Three-hundred microlitres of plasma were used to quantify dihydroceramides, ceramides, sphingomyelins and sphingosine content. The lipid subspecies were extracted and analysed by Liquid Chromatography Mass Spectrometry (LC-MS/MS), at the Lipidomic Core Facility of the University of Bourgogne (Dijon, France).
- Correlation between sphingolipids species concentrations and insulin resistance (HOMA-IR) | Samples taken in 1 single time in the morning, patients fast for 12 hours, on 1 single day
  Three-hundred microlitres of plasma were used to quantify dihydroceramides, ceramides, sphingomyelins and sphingosine content. The lipid subspecies were extracted and analysed by Liquid Chromatography Mass Spectrometry (LC-MS/MS), at the Lipidomic Core Facility of the University of Bourgogne (Dijon, France).
- Correlation between sphingolipids species concentrations and microvascular complications (history of retinopathy, nephropathy and neuropathy) | Samples taken in 1 single time in the morning, patients fast for 12 hours, on 1 single day
  Three-hundred microlitres of plasma were used to quantify dihydroceramides, ceramides, sphingomyelins and sphingosine content. The lipid subspecies were extracted and analysed by Liquid Chromatography Mass Spectrometry (LC-MS/MS), at the Lipidomic Core Facility of the University of Bourgogne (Dijon, France).
- Correlation between sphingolipids species concentrations and macrovascular complications (cardiovascular disease history) | Samples taken in 1 single time in the morning, patients fast for 12 hours, on 1 single day
  Three-hundred microlitres of plasma were used to quantify dihydroceramides, ceramides, sphingomyelins and sphingosine content. The lipid subspecies were extracted and analysed by Liquid Chromatography Mass Spectrometry (LC-MS/MS), at the Lipidomic Core Facility of the University of Bourgogne (Dijon, France).

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided